CLINICAL TRIAL: NCT03787043
Title: A Randomized, Open-label, Single-dosing, 2X2 Crossover Study to Evaluate the Effect of Food on the Safety and Pharmacokinetics of Fixed-dose Combination of MP-513 10mg and Metformin XR 750mg in Healthy Male Volunteers
Brief Title: A Study to Evaluate the Effect of Food on Fixed-Dose Combination of MP-513 10 mg and Metformin XR 750 mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MP_C102
Record Dates: First submitted 2015-10-05; First posted 2018-12-26 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Healthy Volunteers
Keywords: Food Effect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence Group A (Experimental): 1. 1st period: FDC(MP-513 10mg/Metformin XR 750mg) under fasted
  2. 2nd period: FDC(MP-513 10mg/Metformin XR 750mg) under fed
  Interventions: Drug: FDC(MP-513 10mg/Metformin XR 750mg)
- Sequence Group B (Experimental): 1. 1st period: FDC(MP-513 10mg/Metformin XR 750mg) under fed
  2. 2nd period: FDC(MP-513 10mg/Metformin XR 750mg) under fasted
  Interventions: Drug: FDC(MP-513 10mg/Metformin XR 750mg)

INTERVENTIONS:
Drug: FDC(MP-513 10mg/Metformin XR 750mg)
  Other Names: HL1511

SUMMARY:
The purpose of this study is to compare the safety and pharmacokinetic characteristics of fixed-dose combination of MP-513 10mg and metformin XR 750mg administered in a high fat fed state versus fasting state to healthy male volunteers.

DETAILED DESCRIPTION:
1. Randomized, open-label, single-dosing, two-treatment, two-sequence, two-period, crossover design
2. Wash-out period: 14 days from the first dosing
3. Drug concentration analytical device: UPLC-MS/MS

ELIGIBILITY:
Inclusion Criteria:

* A healthy male adult at the age of 20 to 45 (both inclusive) at the time of screening test.
* Body weight equal to or greater than 55 kg and calculated ideal body weight (IBW) within ±20%
* An individual who has been given and fully understood detailed explanations about this study, decides to participate in the study of his own will, and provides written informed consent to comply with instructions.

Exclusion Criteria:

* History or presence of any clinically significant diseases in the hepatobiliary, renal, nervous(central or peripheral), respiratory, hemato-oncology, cardiovascular, urinary, musculoskeletal, immune, ear, nose and throat (ENT), mental, and, particularly, endocrine systems (e.g., diabetes mellitus, hyperlipidemia, etc.).
* History of any gastrointestinal disease that may affect absorption of the study drug (Crohn's disease, ulcer, acute or chronic pancreatitis, etc.) or gastrointestinal surgeries (except for simple appendectomy or hernia repair).
* Hypersensitivity to MP-513 or drugs containing metformin or other drugs in the same class as ingredients or to other drugs
* Vital signs in a sitting position corresponding to at least one of the following criteria: systolic blood pressure ≥ 140 mmHg or < 90 mmHg, or diastolic blood pressure ≥ 95 mmHg or < 60 mmHg.
* Serum creatine > upper limit of reference range
* Required to refrain from food intake for at least 24 hours during the study period due to surgery or religious reason.
* History or presence of drug abuse.
* Administration of drugs that either induce or inhibit drug metabolizing enzymes, such as barbitals, within 1 month prior to the first dosing.
* Intake of food or beverage containing grapefruit or cranberry within 1 week prior to the first dosing.
* Administration of any ethical drugs or traditional Korean herbal medicines within 2 weeks or any over-the-counter drugs or vitamin products within 1 week prior to the first dosing
* An individual who participated in another clinical trial and was administered any investigational product within 3 months prior to the first dosing.
* Whole blood donation within 2 months, apheresis donation within 1 month, or blood transfusion within 1 month prior to the first dosing.
* An individual who drinks excessive amounts of alcohol or who cannot stop drinking alcohol from 24 hours prior to hospital admission through to hospital discharge.
* Having smoked 10 cigarettes/day or more on average over the past 3 months.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
AUC of MP-513 and metformin | 0(pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hours post-dose for each period(a total of 36 times, with 18 times per period)
  PK
Cmax of MP-513 and metformin | 0(pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 36, 48, 72 hours post-dose for each period(a total of 36 times, with 18 times per period)
  PK

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical trials center of Chungnam National University Hospital, Daejeon, Jung-gu, South Korea

IPD SHARING:
Plan to Share IPD: Yes